CLINICAL TRIAL: NCT05138380
Title: Hip Osteoarthritis and Foot Orthoses Trial (HOOT): A Randomized Feasibility Trial
Brief Title: Hip Osteoarthritis and Foot Orthoses Trial (HOOT)
Acronym: HOOT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: La Trobe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HOOT
Record Dates: First submitted 2021-11-02; First posted 2021-12-01 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-03

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Foot Orthoses

STUDY DESIGN:
Intervention Model Description: Two-arm, participant blinded, parallel group feasibility RCT
Who Masked: Participant, Outcomes Assessor
Masking Description: Assessor blinding: Participants complete their own outcome measures (questionnaires) online and are thus not blind. Accelerometry data will be assessor blinded. All outcome measures will be analysed by an investigator blind to participant group allocation. Participants will be instructed not to divulge any aspect of their intervention to the research assistant conducting follow-up assessments.
  Participant blinding: Participants will be advised that they have an equal chance of being allocated to the either shoe insert, and thus are blind to allocation. Participants will also be blind to the study hypothesis, so they are unaware which of the interventions is 'active'.
  Physiotherapist blinding: It is not possible to blind the trial physiotherapist to group allocation. Trial Physiotherapists will however not be involved in assessment of outcome measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foot orthoses (Experimental)
  Interventions: Device: Foot orthoses
- Flat shoe insert (Sham Comparator)
  Interventions: Device: Flat shoe insert

INTERVENTIONS:
Device: Foot orthoses — Manufacturer: Foot Science International.
  Material: High grade thermoformable closed-cell polyolefin foam (medium density)
  Arch support: inbuilt.
  Covering: fabric
  Provided by: Study Practitioner: Registered physiotherapist > 2 years musculoskeletal experience will be trained to prescribe the insert according to the prescription algorithm.
  Where: Administered via telehealth
  When and how much: Week 0 to 1: one telehealth session with study practitioner to fit one pair of pre-fabricated orthoses Week 1 to 2: Follow-up session for questions if required
  Tailoring: Orthoses are fit to comfort. Lengths (S, S, M, L, XL, XXL) (dependent on participant's shoe size). Hardness = Medium density. Modifications: can be cut to size to assist in fit using the shoes original sock liner as a guide, by participants using standard scissors. Heat molding: optional.
  Adherence: Adherence recorded with diary/ log book (insert wear time)
  Other Names: Foot Science International Ltd; Formthotic
  Arms: Foot orthoses
Device: Flat shoe insert — Manufacturer: Foot Science International.
  Material: High grade thermoformable closed-cell polyolefin foam (medium density)
  Arch support: no.
  Covering: fabric
  Provided by: Study Practitioner: Registered physiotherapist > 2 years musculoskeletal experience will be trained to prescribe the insert according to the prescription algorithm.
  Where: Administered via telehealth
  When and how much: Week 0 to 1: one telehealth session with study practitioner to fit one pair of pre-fabricated orthoses Week 1 to 2: Follow-up session for questions if required
  Tailoring: Fit to comfort. Lengths (S, S, M, L, XL, XXL) (dependent on participant's shoe size). Hardness = Medium density. Modifications: can be cut to size to assist in fit using the shoes original sock liner as a guide, by participants using standard scissors. Heat molding: optional.
  Adherence: Adherence recorded with diary/ log book (insert wear time)
  Arms: Flat shoe insert

SUMMARY:
This trial is a randomized feasibility trial to determine the feasibility of comparing two different shoe inserts and on pain, quality of life and physical activity associated with hip osteoarthritis.

DETAILED DESCRIPTION:
Participants will be randomized to one of two groups - contoured prefabricated foot orthoses or flat shoe inserts (the comparator). Participants will be asked to use the inserts daily for a six week period. Adherence to the intervention will be monitored using a daily diary, as well as adverse events and co-interventions. The primary outcome is feasibility domains (Demand, Implementation, Acceptability, Practicality) with secondary outcomes of change in hip-related pain and quality of life and physical activity levels. The primary time-point will be 6-weeks.

ELIGIBILITY:
Inclusion Criteria:

Primary symptomatic and radiographic hip OA, in accordance with the American College of Rheumatology

(i) aged > 45 years;

(ii) pain in the hip or groin for more than 3 months;

(iii) average pain intensity over the past week of > 3 out of 10 (Numerical Rating Scale) during functional tasks like walking, climbing stairs or climbing in/out of a car;

(iv) radiographic confirmation of hip osteoarthritis with a Kellgren-Lawrence score ≥ 2 within the last 12 months;

(v) mild to moderate disability indicated by;

1. able to reciprocally ascend and descend 10 stairs unaided,
2. able to safely walk one city block, and
3. able to jog five meters if required

Exclusion Criteria:

(i) other musculoskeletal lower limb or back conditions requiring assessment or treatment by a health professional (Doctor, Physiotherapist, Podiatrist etc) in the last 6 months;

(ii) have received active treatment for their hip pain by a health professional (eg physiotherapist) in the last 3 months;

(iii) history of hip trauma or surgery on the affected side;

(iv) corticosteroid use (oral or intra-articular injection) in the past 3 months

(v) neurological impairment or condition affecting lower limb function

(vi) conditions or factors affecting ability to take part in the intervention, e.g., unavailable for a 6 week intervention period, routine use of gait aids, uncontrolled hypertension, or morbid obesity (body mass index > 40);

(vii) Use of foot orthoses in the previous 12 months

(viii) systemic inflammatory disease (e.g. rheumatoid arthritis);

(ix) unable to write, read or comprehend English.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-10-26 (Estimated)

PRIMARY OUTCOMES:
Feasibility: adherence | 6 weeks
  Recruitment rate (average 1 participant per week); 50% log-book completion rate (daily); drop-out <20%; 35 hours per week adherence to intervention (log book)

SECONDARY OUTCOMES:
Hip-related pain | Baseline and 6 weeks
  Hip osteoarthritis outcome score: pain sub-scale (HOOS-12). Scores range for 0 (better outcomes) - 100 (worse outcomes)
Hip-related physical function | Baseline and 6 weeks
  Hip osteoarthritis outcome score: function and daily living subscale. Scores range for 0 (better outcomes) - 100 (worse outcomes)
Hip-related quality of life | Baseline and 6 weeks
  hip osteoarthritis outcome score: quality of life subscale: Scores range for 0 (better outcomes) - 100 (worse outcomes)
Fear of movement | Baseline and 6 weeks
  Brief Fear of Movement Scale for osteoarthritis (BFOM); 0 to 24, with a higher score indicating lower fear of movement (better score)
Depressive symptoms | Baseline and 6 weeks
  Patient Health Questionnaire -9: Scored from 0 to 27, participants can be classified as having mild (≥ 5), moderate (≥ 10), moderately severe (≥ 15) and severe (≥ 20) depressive symptoms.
Physical activity- Self-reported | Baseline and 6 weeks
  The International Physical Activity Questionnaire: Participants will be asked to recall their physical activity over the last 7 days with regard to vigorous physical activity, moderate physical activity, walking and sitting.
Physical activity- Walking based physical activity | Baseline and 6 weeks
  Will be measured with a tri-axial accelerometer-based activity monitor that is attached on the thigh (activPAL model 4 micro; PAL Technologies Ltd, Glasgow, UK) and will be expressed as a) daily minutes of moderate and vigorous physical activity using the established 100 steps/minute threshold and b) total daily steps (which captures both inside and outside the home walking activity).
Global rating of change- Physical activity | Week 6
  Seven point rating scale. Much better, better, a little better, no change, a little worse, worse, much worse
Global rating of change- Symptoms | Week 6
  Seven point rating scale. Much better, better, a little better, no change, a little worse, worse, much worse

CONTACTS AND LOCATIONS:
Overall Officials: Adam Semciw, PhD, Principal Investigator — La Trobe University
Locations (1):
- La Trobe University, Bundoora, Victoria, Australia

REFERENCES:
- [Derived] King MG, Hon R, Roughead E, Kemp JL, Pizzari T, Wong J, Menz HB, Taylor NF, Harms A, McClelland JA, Semciw AI. Prefabricated contoured foot orthoses to reduce pain and increase physical activity in people with hip osteoarthritis: A randomised feasibility trial. Physiother Res Int. 2024 Oct;29(4):e2118. doi: 10.1002/pri.2118. PMID 39132922
- [Derived] King MG, Kemp JL, Hon R, Pizzari T, Wong J, Menz H, Taylor NF, Harms A, McClelland JA, Semciw AI. Prefabricated contoured foot orthoses to reduce pain and increase physical activity in people with hip osteoarthritis: protocol for a randomised feasibility trial. BMJ Open. 2022 Sep 6;12(9):e062954. doi: 10.1136/bmjopen-2022-062954. PMID 36691129